CLINICAL TRIAL: NCT03255850
Title: The Impact of Congenital Heart Disease on the Psychological Well Being and Quality of Life in the Hong Kong Chinese Adolescents
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: MPhil_2
Record Dates: First submitted 2017-08-17; First posted 2017-08-21 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Congenital Heart Disease
Keywords: adolescents; quality of life; psychological well-being
MeSH Terms: conditions — Heart Defects, Congenital; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adolescents with CHD: Adolescents with CHD are required to complete the Chinese version of Pediatric Quality of Life Inventory 4.0 Generic Core Scales (PedsQL), Center for Epidemiological Studies -Depression Scale (CES-DC) and Rosenberg Self-Esteem Scale (RSES)
- Healthy control: Data of healthy control who completed the Chinese version of Pediatric Quality of Life Inventory 4.0 Generic Core Scales (PedsQL), Center for Epidemiological Studies -Depression Scale (CES-DC) and Rosenberg Self-Esteem Scale (RSES) are retrieved from previous studies.
- Childhood cancer survivors: Data of childhood cancer survivors who completed the Chinese version of Pediatric Quality of Life Inventory 4.0 Generic Core Scales (PedsQL), Center for Epidemiological Studies -Depression Scale (CES-DC) and Rosenberg Self-Esteem Scale (RSES) are retrieved from previous studies.

SUMMARY:
This study aims to examine the psychological well-being and QoL of Hong Kong Chinese adolescents with CHD by

* comparing the self-esteem level, depressive symptoms, and quality of life of adolescents suffering from CHD with healthy norms and cancer survivors.
* identifying possible factors affecting the quality of life of adolescents suffering from CHD.

DETAILED DESCRIPTION:
Congenital heart disease (CHD) is the most common type of congenital malformation in the world with birth prevalence as 8 per 1000 live births. Survival rate has been drastically improved as a result of improvement in surgical treatments and intensive care but adolescents with CHD still suffer from limitations on their psychological functioning and restrained quality of life. Number of evidences have indicated that adolescents with CHD experience more depressive symptoms and lower self-esteem level than their healthy counterparts. In addition, adolescents with CHD are more prone to develop emotional and behavioral problems than their healthy norms. Given the above issues, It is imperative for nurses to develop psychological interventions to promote psychological well-being among adolescents with CHD, with the goal of improving their quality of life. There have been increasing concerns worldwide on the quality of life of such population especially on how does the disease pose threats on their daily living. However, at present, there is no study examining how does CHD affect the psychological well-being and quality of life in Hong Kong Chinese adolescents. It is explicit that Hong Kong has a distinctively different cultural context from that of the West. Hence, the effects of CHD and its treatments are likely to differ markedly in the two regions .To conclude, results of previous studies from the West may not fit into Hong Kong Chinese cultural context.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients with congenital heart disease
* aged at 12-17 years old
* fluent in Cantonese and able to read Chinese

Exclusion Criteria:

* pediatrics with major developmental delay or having significant co-morbid medical condition
* visiting because of altering in clinical condition
* having acquired heart disease or non-structural heart disease

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric with congenital heart disease, aged at 12-17 years old, fluent in Cantonese and are attending the day centre and specialized outpatient sector of Department of Pediatric Cardiology in Queen Mary Hospital .
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Health related quality of life | 1 day
  Quality of life is measured by Pediatric Quality of Life Inventory 4.0 Generic Core Scales (PedsQL) which aims at measuring patient's perceptions of the patient's HRQOL in various aspects namely the impact of disease and treatment on an individual's physical functioning(8 items ), emotional functioning(5 items), social functioning(5 items), and school functioning(5 items). The 5-point Likert scale is used for indicating the frequency of a problem has been during the past one month ,0=never a problem, 1=almost never a problem, 2=sometimes a problem, 3=often a problem and 4=almost always a problem. The PedsQL core scales can be completed within 10-15 minutes. Reversed scoring will be used to evaluate the items and linear transformed into 0-100 scale, thus higher PedsQL scores represents greater HRQOL.

SECONDARY OUTCOMES:
Self-esteem | 1-day
  Self-esteem level is measured by the Rosenberg Self-Esteem Scale (RSES). It consists of
Depressive symptoms | 1-day
  Depressive symptoms is measured by The Center for Epidemiologic Studies Depression Scale

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] So SCY, Li WHC, Ho KY. The impact of congenital heart disease on the psychological well-being and quality of life of Hong Kong Chinese adolescents: A cross-sectional study. J Clin Nurs. 2019 Sep;28(17-18):3158-3167. doi: 10.1111/jocn.14864. Epub 2019 Apr 21. PMID 30938874